CLINICAL TRIAL: NCT00663104
Title: Effect of Exercise and Exercise + Phytoestrogen on Bone, Metabolic Syndrome Criteria and Complaints of the Early Menopause
Brief Title: Effect of Exercise and Phytoestrogen on Bone, Metabolic Syndrome Criteria and Complaints of the Early Menopause
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Siemens-Betriebskrankenkasse (Industry)
Responsible Party: Principal Investigator, Wolfgang Kemmler, Principal Investigator, University of Erlangen-Nürnberg Medical School
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: OFZ-Trace
Record Dates: First submitted 2008-04-21; First posted 2008-04-22 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Bone Diseases; Metabolic Syndrome X; Coronary Disease
Keywords: early menopause; exercise; phytoestrogen; bone; CHD-risk factors
MeSH Terms: conditions — Bone Diseases; Metabolic Syndrome; Coronary Disease; Primary Ovarian Insufficiency; Motor Activity | interventions — Exercise; black cohosh root extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): exercise (3 sessions/week)
  Interventions: Behavioral: exercise
- 2 (Active Comparator): exercise and "phytoestrogen" (cimicifuga racemosa)
  Interventions: Behavioral: exercise + cimicifuga racemosa
- 3 (Placebo Comparator): wellness control, placebo
  Interventions: Behavioral: wellness control, placebo

INTERVENTIONS:
Behavioral: exercise — exercise: 3 joint sessions/week for 12 months
  Arms: 1
Behavioral: exercise + cimicifuga racemosa — exercise: 3 sessions/week for 12 months,cimicifuga racemosa (40 mg/d)
  Arms: 2
Behavioral: wellness control, placebo — 2x10 weeks with 1 session/week of low volume, low intensity wellness training over 12 months, placebo
  Arms: 3

SUMMARY:
The aim of the study is to compare the effect of a progressive, periodized exercise training designed to impact bone, CHD-risk-factors and menopausal complaints versus the combined effect of exercise and "phytoestrogen" (cimicifuga racemosa; CR). After randomization, 84 females 1-3 year postmenopausal with no medication or illness affecting bone metabolism exercise over 12 months (EG; 42 with, 42 without CR), 42 women serve as wellness-control. Three group training sessions/week will be performed in the EG. Both groups will be individually supplemented with calcium and Vit-D (cholecalciferol).

ELIGIBILITY:
Inclusion Criteria:

* 1-3 years early postmenopausal
* Caucasian race

Exclusion Criteria:

* CHD-diseases
* thrombosis, embolism
* fractures at lumbar spine or hip
* secondary osteoporosis
* hyperparathyroidism
* medication, diseases with impact on muscle or bone
* cancer and hormone derived malign diseases
* weight reduction of > 5 kg during the last 6 months

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2008-04; Primary Completion 2009-06 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density | baseline, 12 month

SECONDARY OUTCOMES:
body composition | baseline, 12 month
blood lipids, glucose | baseline, 12 month
blood pressure | baseline, 12 month
10 year CHD-risk | baseline, 12 months
menopausal complaints | baseline, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bebenek, MS, Principal Investigator — University of Erlangen-Nürnberg Medical School; Wolfgang Kemmler, PhD, Study Director — University of Erlangen-Nürnberg Medical School; Willi A Kalender, Professor, PhD, Study Chair — University of Erlangen-Nürnberg Medical School
Locations (1):
- Institute of Medical Physics, Erlangen, Germany

REFERENCES:
- [Background] Kemmler W, Lauber D, Weineck J, Hensen J, Kalender W, Engelke K. Benefits of 2 years of intense exercise on bone density, physical fitness, and blood lipids in early postmenopausal osteopenic women: results of the Erlangen Fitness Osteoporosis Prevention Study (EFOPS). Arch Intern Med. 2004 May 24;164(10):1084-91. doi: 10.1001/archinte.164.10.1084. PMID 15159265
- [Background] von Stengel S, Kemmler W, Kalender WA, Engelke K, Lauber D. Differential effects of strength versus power training on bone mineral density in postmenopausal women: a 2-year longitudinal study. Br J Sports Med. 2007 Oct;41(10):649-55; discussion 655. doi: 10.1136/bjsm.2006.033480. Epub 2007 Jun 5. PMID 17550916
- [Background] Kemmler W, von Stengel S, Weineck J, Lauber D, Kalender W, Engelke K. Exercise effects on menopausal risk factors of early postmenopausal women: 3-yr Erlangen fitness osteoporosis prevention study results. Med Sci Sports Exerc. 2005 Feb;37(2):194-203. doi: 10.1249/01.mss.0000152678.20239.76. PMID 15692313